CLINICAL TRIAL: NCT05963464
Title: RADIOSO MILAN I (RADar Reflector localisatiOn-SCOUT for carcinOma Mammae, the MILAN IEO Experience I)
Acronym: RADIOSO
Status: Recruiting | Type: Observational
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: IEO 1911/
Record Dates: First submitted 2023-07-19; First posted 2023-07-27 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-07

CONDITIONS: Breast Cancer; Occult Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: SCOUT® Radar occult breast lesion Localization — The SCOUT® Radar occult breast lesion Localization (SRL) uses non-radioactive micro-impulses to guide surgical excision in real time.

SUMMARY:
This is a monocentric prospective observational study for patients with clinical undetectable breast lesions and indications to breast conserving surgery for histological characterization.

The SCOUT® Radar occult breast lesion Localization (SRL) consists of an implantable reflector, a detector handpiece and a console and it uses non-radioactive micro-impulses to guide surgical excision in real time.

The study describes the experience with 300 patients at the European Institute of Oncology.

The primary endpoints of the study are the rates of successful positioning, localization and recovery of the reflector SRL.

DETAILED DESCRIPTION:
It has been estimated that 31,8% of breast cancer patients undergo pre-operational lesion localization. Of them, 19% have been previously administered neoadjuvant chemotherapy (NACT). Based on retrospective data, NACT administration is believed to steadily increase by 1,3%, each year.

The IEO Breast Division Program aims at improving the treatment and planning options available to patients referred for radio guided breast surgery.

At IEO, ROLL remains the standard of care. From its inception 25 year ago to the present day,the investigators have gained significant expertise and now perform more than 1000 procedures per year.

The investigators believe that SRL (SCOUT® Radar occult breast lesion Localization) could be added to the procedure of reference in the following cases, still under investigation, where it seems to present some advantages when compared to ROLL:

1. Long-term positioning of the reflector, as in the case of patients undergoing neoadjuvant treatment
2. Reflector placement in malignant lymphadenopathy prior to neoadjuvant chemotherapy
3. Placement of multiple reflectors, or use of both SRL and ROLL in patients with multifocal or multicentric neoplasia referred for conservative surgery
4. BI-RADS 5 patients suspected for ductal carcinoma in situ (DCIS) and eligible for conservative surgery, could undergo reflector placement after vacuum-assisted breast biopsy (VABB) and also be scheduled for Monday morning surgery
5. Placement of the reflector using MR-compatible introducer needles

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of nonpalpable breast or lymph nodes
* Patients referred to IEO for breast surgery
* Patients between 18 and 90 years old
* Female patients
* Conservative surgery
* Patients willing and able to follow the study procedures and available for follow-up over the entire duration of the study

Exclusion Criteria:

* Patients known or suspected to be allergic to materials similar to those in the SAVI SCOUT components (nickel)
* Any condition that may expose the individual to a higher risk or preclude the study from achieving full compliance or completion.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosis of nonpalpable breast lesion or lymph nodes requiring conservative surgical excision.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of successful positioning of the reflector | 1 week
  Percentage of reflectors successfull positioned
Rate of successful localization of the reflector | 6 months
  Percentage of reflectors successfull localized
Rate of successful recovery of the reflector | 6 months
  Percentage of reflectors successfull recovered

SECONDARY OUTCOMES:
Rate of cases with negative margins | 6 months
  percentage of cases with negative margins
Rate of cases that have required a second excision | 6 months
  Percentage of cases that have required a second excision

CONTACTS AND LOCATIONS:
Overall Officials: Gianmatteo Pagani, MD, Principal Investigator — European Institute of Oncology
Locations (1):
- European Institute of Oncology, Milan, Italy

IPD SHARING:
Plan to Share IPD: No